CLINICAL TRIAL: NCT05991362
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose and Multiple-dose Study Evaluating the Pharmacokinetics and Safety of GFH312 in Healthy Chinese Subjects
Brief Title: A Phase I Study of GFH312 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Genfleet Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFH312X1102
Record Dates: First submitted 2023-07-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD:100mg (Experimental): Participants received single PO dose of GFH312 100 mg.
  Interventions: Drug: GFH312 100 mg
- SAD:200mg (Experimental): Participants received single PO dose of GFH312 200 mg.
  Interventions: Drug: GFH312 200 mg
- MAD:120mg (Experimental): Participants received multiple PO doses of GFH312 120 mg for 14 days.
  Interventions: Drug: GFH312 120mg
- Placebo (Placebo Comparator): Participants receiving placebo matching with the GFH312 dose groups
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GFH312 100 mg — Participants receive single dose of GFH312 100 mg orally
  Other Names: GFH312
  Arms: SAD:100mg
Drug: GFH312 200 mg — Participants receive single dose of GFH312 200 mg orally
  Other Names: GFH312
  Arms: SAD:200mg
Drug: GFH312 120mg — Participants receive daily dose of GFH312 120mg orally for fourteen consecutive days
  Other Names: GFH312
  Arms: MAD:120mg
Other: Placebo — Participants receive placebo matching with GFH312
  Arms: Placebo

SUMMARY:
The aim of this study was to evaluate the pharmacokinetic profile and observe the safety of GFH312 after single and multiple administrations in healthy Chinese subjects.

DETAILED DESCRIPTION:
This study was planned to enroll about 26 healthy subjects, subjects were planned to receive single administration of 100 mg GFH312, single administration of 200 mg GFH312, or multiple administrations of 120 mg GFH312, as well as their matching placebo. Subjects were randomized in 3:1 ratio in the single dose cohorts and in 4:1 ratio in the multiple dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent;
* Male or female healthy subjects aged 18-55 years (inclusive) (single sex ratio not less than 25% of the sample size of each cohort);
* Body mass index (BMI) between 18-28 kg/m2 (inclusive), and weight ≥ 50kg; BMI = Weight (kg) /[Height (m)]2.
* During the screening period and day 1, patients with normal or abnormal results but no clinical significance based on detailed medical history, comprehensive physical examination, laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function), 12-lead electrocardiogram and vital signs.
* Able to communicate well with researchers, understand and comply with research requirements.

Exclusion Criteria:

* Any procedure or disease that may significantly alter drug absorption, distribution, metabolism, or excretion, or participation in this study may compromise the safety of the subject.
* Tuberculin test positive
* Abnormal electrocardiogram with clinical significance
* Use any prescription drugs, Chinese herbs and/or OTC or health products within 2 weeks before starting the administration.
* Women who are pregnant or breastfeeding, or subjects with positive pregnancy test results at the time of screening or at baseline, or who plan to become pregnant during the study period or within 30 days after the end of the study.
* Subjects who have any factors deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4.
  The maximum observed plasma concentration (Cmax) was estimated based on the plasma concentrations of GFH312.
Time to peak drug concentration (Tmax) of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4.
  The time it takes for a drug to reach the maximum concentration (Cmax) after administration of GFH312
Terminal Elimination Half Life (t1/2) of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4; for multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  The terminal elimination half-life (t1/2) was estimated based on the plasma concentrations of GFH312
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4.
  The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) was estimated based on the plasma concentrations of GFH312
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4.
  The area under the plasma concentration-time curve from time zero to infinity (AUC 0-inf) was estimated based on the plasma concentrations of GFH312
The apparent systemic (or total body) clearance from plasma (or serum or blood (CL/F) following extravascular administration of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4; for multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  The systemic clearance (CL) was estimated based on the plasma concentrations of GFH312
The apparent volume of distribution during the terminal elimination phase (Vd/F) following extravascular administration of GFH312 | For single dose groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 6, 8, 12 hours on day1; day2, day3, day4; for multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  The volume of distribution was estimated based on the plasma concentrations of GFH312
The observed maximum plasma (or serum or blood) concentration following drug administration at steady state (Cmax,ss) | For multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  Observed maximum concentration in the dosing interval at steady state
The lowest plasma (or serum or blood) concentration observed during a dosing interval at steady state (Cmin,ss) | For multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  Observed minimum concentration in the dosing interval at steady state.
Time to reach maximum concentration in the dosing interval at steady state (Tmax,ss) | For multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  If the same Cmax concentration occurs at different time points, Tmax is assigned to the first occurrence of Cmax.
The area under the plasma (or serum or blood) concentration-time curve from time zero to the end of the dosing interval tau (AUCtau,ss) | For multiple doses groups 30 minutes pre-dose, and at 0.5, 1, 2, 4, 8, 12 hours on day 1; day2, day7, day 13, day14, day15.
  Dose-normalized AUC0- τ, calculated as AUC0-τ divided by actual dose administered.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | up to 30 days after the last study drug administration
  An adverse event (AE) is any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly or birth defect in the offspring of a participant who received the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: LU Yongning, PHD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No